CLINICAL TRIAL: NCT00258687
Title: A Phase I Trial of Vaccination With Autologous, Lethally Irradiated Tumor Cells Engineered by Adenoviral Mediated Gene Transfer to Secrete Granulocyte-Macrophage Colony Stimulating Factor in Pediatric and Adult Patients
Brief Title: Vaccine Trial for Clear Cell Sarcoma, Pediatric Renal Cell Carcinoma, Alveolar Soft Part Sarcoma and Children With Stage IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, F. Stephen Hodi, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-115
Record Dates: First submitted 2005-11-23; First posted 2005-11-28 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Sarcoma, Clear Cell; Sarcoma, Alveolar Soft Part; Renal Cell Carcinoma; Melanoma
Keywords: GVAX; GM-CSF; Adenoviral mediated gene transfer; Pediatric Melanoma
MeSH Terms: conditions — Sarcoma, Clear Cell; Sarcoma, Alveolar Soft Part; Carcinoma, Renal Cell; Melanoma

ARMS (2):
- Treatment Arm A (Experimental): GVAX for Sarcoma / Renal Cell Patients
  Interventions: Biological: GVAX
- Treatment Arm B (Experimental): GVAX for Pediatric Melanoma Patients
  Interventions: Biological: GVAX

INTERVENTIONS:
Biological: GVAX — 4 vaccines every two weeks

SUMMARY:
The purpose of this study is to learn if a vaccine made from the patient's own tumor cells, then genetically modified to secrete granulocyte-macrophage colony-stimulating factor (GM-CSF), will delay or stop the growth of the tumor. It will also look at the vaccine's effects on the immune system and the side effects of giving a vaccine made from a subject's own cancer cells.

DETAILED DESCRIPTION:
The patient will have surgery to remove a portion of the tumor. This tumor is then brought to a special, certified laboratory where it is broken up into single cells and then washed.

Specially trained laboratory technicians then use a method known as adenoviral mediated gene transfer, which adds a new gene to the cancer calls. This gene causes the cells to make GM-CSF, a powerful hormone that stimulates the immune system. The cells are then given enough radiation so that they will never grow, but not enough to completely destroy them, developing a vaccine.

The patient is then injected with the vaccine on days 0, 7, 14, 28, and then every two weeks until the supply of vaccine has run out. The amount of vaccine that can be made depends upon the total amount of cells taken from the tumor. The actual injections are like childhood vaccinations that go under the skin or into muscle and a different place will be used for each injection.

It is hoped that the cancer cells that have been made to secrete the hormone GM-CSF will cause the patient's immune system to attack the cancer in other parts of the body.

If the tumor yields enough cells, the patient will also be given an injection of non-transduced irradiated tumor cells. Non-transduced means that the gene for GM-CSF has not been added to these cells as it has for the vaccines. This is done to measure the amount of reaction of the immune system caused by the vaccine. This injection is measuring delayed type hypersensitivity, or DTH.

The patient will be asked to undergo optional skin biopsies of the vaccine and DTH sites to see if an immune reaction is occuring at the injection sites 2 days after vaccine 1 and vaccine 5.

The following tests and procedures will be performed through out the study: physical exam, blood samples, immune studies, vital signs and physical exam.

At week 10 in the patient's treatment, or earlier if the doctor feels it is necessary, the patient will undergo a chest, abdomen and pelvic XT scan. A brain MRI will be performed if there were any abnormalities on the first brain MRI or if any new central nervous system symptoms have developed.

If the patient's disease has not disappeared or if new lesions have been found after the patient receives at least six vaccines, they may have the opportunity to undergo a second course of study treatment.

Patients may participate in this study until one of the following happens: All vaccine created from the tumor has been given to the patient; the patient's disease worsens; the patient experiences an unacceptable and/or harmful side effect; the patient becomes pregnant; the patient is unable to follow the study plan; or the patient's doctor feels it is no longer in the best interest of the patient to continue.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0 or 1
* Estimated life expectancy of greater than 6 months
* Greater than or equal to 4 weeks from chemotherapy, radiotherapy, immunotherapy, or systemic glucocorticoid therapy
* Greater than or equal to 6 months from prior bone marrow or peripheral blood stem cell (PBSC) transplant
* Histologically confirmed alveolar soft part sarcoma or clear cell sarcoma at any age.
* Evidence of metastatic disease, including having spread either to distant sites that may include brain metastases, or to regional lymph nodes alone, or locally advanced primary lesion that is not fully surgically resectable at study entry.
* Histologically confirmed Stage IV renal cell carcinoma (patients with brain metastases still eligible)
* Any patients with Stage IV renal cell carcinoma under the age of 25 years who do not have a renal cell carcinoma predisposition syndrome
* Patients with Stage IV melanoma and under the age of 18 years

Exclusion Criteria:

* Uncontrolled active infection
* Pregnancy or nursing mothers
* Infection with HIV, hepatitis B or hepatitis C
* Any other significant medical, surgical, or psychiatric condition that may interfere with compliance with protocol regimen
* Other current malignancies apart from any in situ cancer or basal or squamous cell carcinoma
* Pediatric melanoma only: infants with transplacentally acquired melanoma; or children with brain metastases and malignant melanoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2006-07 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
To determine the safety and feasibility of preparation and administration of vaccine in patients with metastatic or locally advanced clear cell sarcoma (CCS), alveolar soft part sarcoma (ASPS) and translocation associated renal cell carcinoma (RCC) | Years

SECONDARY OUTCOMES:
To determine the disease response, immune response, and overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: F. Stephen Hodi, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Children's Hospital Boston, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Background] Soiffer R, Hodi FS, Haluska F, Jung K, Gillessen S, Singer S, Tanabe K, Duda R, Mentzer S, Jaklitsch M, Bueno R, Clift S, Hardy S, Neuberg D, Mulligan R, Webb I, Mihm M, Dranoff G. Vaccination with irradiated, autologous melanoma cells engineered to secrete granulocyte-macrophage colony-stimulating factor by adenoviral-mediated gene transfer augments antitumor immunity in patients with metastatic melanoma. J Clin Oncol. 2003 Sep 1;21(17):3343-50. doi: 10.1200/JCO.2003.07.005. PMID 12947071
- [Background] Salgia R, Lynch T, Skarin A, Lucca J, Lynch C, Jung K, Hodi FS, Jaklitsch M, Mentzer S, Swanson S, Lukanich J, Bueno R, Wain J, Mathisen D, Wright C, Fidias P, Donahue D, Clift S, Hardy S, Neuberg D, Mulligan R, Webb I, Sugarbaker D, Mihm M, Dranoff G. Vaccination with irradiated autologous tumor cells engineered to secrete granulocyte-macrophage colony-stimulating factor augments antitumor immunity in some patients with metastatic non-small-cell lung carcinoma. J Clin Oncol. 2003 Feb 15;21(4):624-30. doi: 10.1200/JCO.2003.03.091. PMID 12586798